CLINICAL TRIAL: NCT03901144
Title: A Phase 2 Randomised Controlled Trial of a NOVel Moisturiser for Atopic Dermatitis: Effect on the Skin Barrier in Adults With a Predisposition to a Skin Barrier Defect
Brief Title: A NOVel Moisturiser for Atopic Dermatitis: Effect on the Skin Barrier
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACO Hud Nordic AB (Industry)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Novum ACO-CT-2018-01; 2018-002945-12 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; skin barrier; moisturiser; emollient
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Every patient use three different creams (1 test cream, 2 reference creams) and one untreated area. They are their own controls
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test cream (2% urea/20% glycerol) (Experimental): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Interventions: Drug: 2% urea/20% glycerol cream
- Reference cream 1: Miniderm® 20% cream (20% glycerol) (Active Comparator): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Interventions: Drug: Miniderm® 20% cream
- Reference cream 2: Diprobase® cream (cream without humectants) (Active Comparator): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Interventions: Drug: Diprobase® cream
- Untreated (No Intervention): Untreated skin area on the volar forearm

INTERVENTIONS:
Drug: 2% urea/20% glycerol cream — Moisturizing cream for topical application
  Other Names: Miniderm Duo 20 mg/g + 200 mg/g cream; Canomini 20 mg/g + 200 mg/g cream
  Arms: Test cream (2% urea/20% glycerol)
Drug: Miniderm® 20% cream — Moisturizing cream for topical application
  Arms: Reference cream 1: Miniderm® 20% cream (20% glycerol)
Drug: Diprobase® cream — Emollient cream for topical application
  Arms: Reference cream 2: Diprobase® cream (cream without humectants)

SUMMARY:
Atopic dermatitis (AD) is among the most common chronic types of inflammatory skin disease and it is characterised by exacerbations or relapses over years. The patients have a genetically impaired skin barrier that can be evaluated by measuring the transepidermal water loss (TEWL), which is increased in both dry skin and clinically normal skin in AD patients. Moisturisers are first line treatment for AD patients and moisturisers are the most prescribed products in dermatology. The use of moisturisers have been found to reduce the need for steroids.

The newly developed moisturizing cream 1107.57 is intended for people with dry skin symptoms, such as dryness, itching, and flaking. As most people with dry skin of different origin have an impaired skin barrier function, it is important to investigate the possible influence on the skin barrier after long-term (several weeks') treatment. It is of utmost importance to evaluate different moisturisers head-to-head in order to facilitate an evidence-based choice of moisturiser.

The primary objective of the trial is to determine whether applying the test cream 1107.57 for 4 weeks is superior in terms of skin barrier strengthening, when compared with (1) no treatment and (2) two reference creams in adults with a predisposition to a skin barrier defect. Secondary objectives are to determine whether there is a difference between 1107.57 and (1) no treatment and (2) the two reference creams in skin moisturization, tolerability, cream consumption and safety.

Participants will treat their lower volar forearms for 28 days with three different creams (test cream and two reference creams) and leave one area untreated as a control. Each forearm will have two different treatment areas and treatment allocation will be randomized. One Finger Tip Unit (FTU) of each cream will be applied twice daily on the designated study area for 28 days. On day 1 and 29 the transepidermal water loss (TEWL) and skin capacitance is measured on their forearms to evaluate the effect on skin barrier function and skin hydration. Furthermore, on day 31, after challenge with 1 % sodium lauryl sulphate (SLS) on day 29, the susceptibility to irritation caused by SLS will be evaluated visually and by measuring TEWL on their forearms. Study participants will attend visits at the start of randomised therapy and on day 5, 15, 29 and 31. During the study period the participants will also grade and evaluate the tolerability of the different creams.

ELIGIBILITY:
Inclusion Criteria:

The participants have to meet all of the following criteria to be eligible to enter the study:

* Willing and able to provide informed consent
* Male or female and aged 18 years or above
* Volunteers able to read and understand English
* A personal history of atopic dermatitis

Exclusion Criteria:

Participants meeting any of the following criteria will not be permitted to enter the study:

* Eczema on the volar forearms requiring anti-inflammatory treatment
* Possible allergy to ingredients in the study medications.
* Any serious current medical condition which, in the opinion of the Investigator, may interfere with the evaluation of the results or may be contraindicated by the use of the test medications
* Use of any concomitant medication that may interfere with the study related activities or assessment of efficacy, as judged by the Investigator
* Use of any topical product, including cosmetic leave-on products on the volar forearms, within 1 week prior to, and throughout the study
* Female participant who, according to the participant, is pregnant or breast-feeding, or plans to become pregnant during the course of the study
* Any participant-related factor suggesting potential poor compliance with study procedures (e.g. psychiatric disorders, history of alcohol or substance abuse), as judged by the Investigator
* Enrolment in any interventional study or use of an investigational drug within 3 months prior to the screening visit
* Volunteers judged by the PI to be inappropriate for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Sheffield Medical School, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Medications prohibited to use >28 Days, 28 Days, 14 Days and 7 Days, respectively, Prior to Baseline/Day 1 and throughout the study are listed in the Clinical Trial Protocol
  Use of bland (non-medicated) emollients, moisturisers or sunscreen on the test areas, within 7 days prior to Visit 1 was also prohibited
  Use of bland (non-medicated) emollient(s) was permitted during the study to manage dry skin in areas surrounding but not on or overlapping the test areas.
Units Other Than Participants: Skin areas
Groups:
- Test Cream (2% Urea/20% Glycerol); Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Reference Cream 2: Diprobase® Cream (Cream Without Humectants): All participants used 3 creams on their lower volar forearms and one area was left untreated. I Finger Tip Unit of each cream was applied every morning and evening for 28 days
- Untreated: All participants used 3 creams on their lower volar forearms and one area was left untreated. No cream was applied on this area
Period: Overall Study
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Started (Each participant used all three creams and had one area untreated, i.e. 4 treatment areas per subject. Total number of subjects was 50) | 50; 50 Skin areas | 50; 50 Skin areas | 50; 50 Skin areas | 50; 50 Skin areas
Completed (Each participant used all three creams and had one area untreated, i.e. 4 treatment areas per subject. Total number of completed subjects was 49) | 49; 49 Skin areas | 49; 49 Skin areas | 49; 49 Skin areas | 49; 49 Skin areas
Not Completed | 1; 1 Skin areas | 1; 1 Skin areas | 1; 1 Skin areas | 1; 1 Skin areas
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Each participant use all three creams and one skin area is untreated. 4 skin areas per subject was evaluated.
Groups:
- Subject Using 3 Creams: Each subject used three creams on their volar forearms and had one skin area untreated 4 treated skin areas: Test cream Glycerol cream Cream without humectants Untreated
Arm/Group | Subject Using 3 Creams
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 49

OUTCOME MEASURES:

1. Primary Outcome: Skin Barrier Strengthening Effect by Measurement of Trans Epidermal Water Loss (TEWL) Before and After Induction of Skin Irritation
Description: The change in TEWL from treated and untreated skin before and after induction of skin irritation with SLS. SLS increases TEWL. An effective treatment protects skin from irritation and less TEWL increase is anticipated compared to untreated skin
Time Frame: day 29 prior to irritant application and day 31 following application
Population: Each participant used three creams on their volar forearms and one skin area was left untreated. A skin irritant was applied on each treatment area (n=4) after end of cream treatment period. The irritant was left on the skin for 24h and the Trans Epidermal Water Loss (TEWL) was measured after another 24h and compared to TEWL measured after treatment but before application of irritant
Measure: Mean (Standard Deviation); unit: TEWL (g/m^2·h) change from day 29 to 31
Units Other Than Participants: skin areas on volar forearms
Groups:
- Test Cream (2% Urea/20% Glycerol): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Test cream: Moisturizing cream for topical application
- Reference Cream 1: Miniderm® 20% Cream (20% Glycerol): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Glycerol cream: Moisturizing cream for topical application
- Reference Cream 2: Diprobase® Cream (Cream Without Humectants): Topical cream, 1 Finger Tip Unit per treatment area on the lower volar forearms twice daily for 28 days
  Cream without humectants: Emollient cream for topical application
- Untreated: Untreated are on the volar forearm
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Number analyzed (Participants) | 49 | 49 | 49 | 49
Number analyzed (skin areas on volar forearms) | 49 | 49 | 49 | 49
TEWL (g/m^2·h) change from day 29 to 31 | 19.790 (13.860) | 24.680 (14.693) | 29.648 (14.299) | 28.646 (13.668)
Statistical Analysis 1: Comparison: Test Cream (2% Urea/20% Glycerol) vs Untreated; Summary of TEWL (g/m2h) change from day 29 to day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -9.026, 95% CI 2-sided [-12.562 to -5.489]
Statistical Analysis 2: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Summary of TEWL (g/m2h) change from day 29 to day 31; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = -4.194, 95% CI 2-sided [-7.760 to -0.629]
Statistical Analysis 3: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 2: Diprobase® Cream (Cream Without Humectants); Summary of TEWL (g/m2h) change from day 29 to day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -9.021, 95% CI 2-sided [-12.602 to -5.440]

2. Primary Outcome: Skin Barrier Strengthening Effect by Measurement of Skin Redness Before and After Induction of Skin Irritation as Assessed by the Erythema Index (Change From Day 29 to Day 31)
Description: Skin redness measurement by Objective Erythema (2D Skin Imaging) on treated and untreated skin before (day 29) and after (day 31) induction of skin irritation with SLS. Captured 2D images are analysed to determine the skin erythema index (degree of redness, arbitrary numerical value), where a higher value denotes a stronger reaction/more redness. An effective treatment is anticipated to protect the skin from irritation, i.e. a weaker reaction from SLS/less redness compared to the untreated skin. Data is presented as change from day 29 to day 31
Time Frame: The 2D Skin Imaging was performed on day 15, day 29 and on day 31. Only day 29 and 31 was included in the statistical analysis
Population: In some participants it was not possible to analyze all images, therefore the Overall Number of Participants Analyzed in this outcome measure differs compared to the total number of participants included in the study
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Units Other Than Participants: skin areas on volar forearms
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Number analyzed (Participants) | 46 | 46 | 45 | 46
Number analyzed (skin areas on volar forearms) | 46 | 46 | 45 | 46
Arbitrary Units | 13.261 (6.9086) | 14.833 (6.0440) | 17.981 (7.3550) | 16.747 (6.7629)
Statistical Analysis 1: Comparison: Test Cream (2% Urea/20% Glycerol) vs Untreated; Summary of Objective Erythema (2D Skin Imaging) change from day 29 to day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.538, 95% CI 2-sided [-5.114 to -1.962]
Statistical Analysis 2: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Summary of Objective Erythema (2D Skin Imaging) change from day 29 to day 31; Test type: Superiority; p = 0.031, ANCOVA; Mean Difference (Final Values) = -1.748, 95% CI 2-sided [-3.332 to -0.164]
Statistical Analysis 3: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 2: Diprobase® Cream (Cream Without Humectants); Summary of Objective Erythema (2D Skin Imaging) change from day 29 to day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.744, 95% CI 2-sided [-6.332 to -3.156]

3. Primary Outcome: Skin Barrier Strengthening Effect by Measurement of Skin Redness Before and After Induction of Skin Irritation as Assessed by Mexameter (Change From Day 29 to Day 31)
Description: Objective skin redness measurement by Mexameter on treated and untreated skin before (day 29) and after (day 31) induction of skin irritation with SLS. Skin redness is measured using a C&K Mexameter probe to quantify SLS-induced skin irritation (arbitrary numerical scale). An effective treatment is anticipated to protect the skin from irritation, i.e. a weaker reaction from SLS/less redness compared to the untreated skin. Data is presented as change from day 29 to day 31
Time Frame: Measured on day 29 and 31
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Units Other Than Participants: skin areas on volar forearms
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Number analyzed (Participants) | 48 | 48 | 47 | 48
Number analyzed (skin areas on volar forearms) | 48 | 48 | 47 | 48
Arbitrary Units | 80.859 (53.901) | 82.893 (53.150) | 106.39 (56.315) | 98.951 (53.917)
Statistical Analysis 1: Comparison: Test Cream (2% Urea/20% Glycerol) vs Untreated; Summary of Redness-Mexameter change from day 29 to day 31; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = -19.077, 95% CI 2-sided [-31.325 to -6.829]
Statistical Analysis 2: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Test type: Superiority; p = 0.471, ANCOVA; Mean Difference (Final Values) = -4.493, 95% CI 2-sided [-16.787 to 7.801]
Statistical Analysis 3: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 2: Diprobase® Cream (Cream Without Humectants); Summary of Redness - Mexameter change from day 29 to day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -27.035, 95% CI 2-sided [-39.372 to -14.698]

4. Primary Outcome: Skin Barrier Strengthening Effect by Measurement of Skin Redness Before Induction of Skin Irritation as Assessed by Visual Scoring
Description: Skin redness by visual scoring on treated and untreated skin before induction of skin irritation with SLS. Skin redness was evaluated on a 4-point visual scale from 0 to 3, where 0 indicates no redness/reaction and 3 indicates strong erythema.
Time Frame: Skin redness was scored on day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: skin areas on volar forearms
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Number analyzed (Participants) | 49 | 49 | 49 | 49
Number analyzed (skin areas on volar forearms) | 49 | 49 | 49 | 49
units on a scale | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Primary Outcome: Skin Barrier Strengthening Effect by Measurement of Skin Redness After Induction of Skin Irritation as Assessed by Visual Scoring
Description: Skin redness by visual scoring on treated and untreated skin after induction of skin irritation with SLS. Skin redness was evaluated on a 4-point visual scale from 0 to 3, where 0 indicates no redness/reaction and 3 indicates strong erythema.
Time Frame: Skin redness was scored on day 31
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: skin areas on volar forearms
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
Number analyzed (Participants) | 49 | 49 | 49 | 49
Number analyzed (skin areas on volar forearms) | 49 | 49 | 49 | 49
units on a scale | 0.99 (0.691) | 1.08 (0.649) | 1.45 (0.718) | 1.35 (0.680)
Statistical Analysis 1: Comparison: Test Cream (2% Urea/20% Glycerol) vs Untreated; Summary of Visual Redness at day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.354, 95% CI 2-sided [-0.558 to -0.150]
Statistical Analysis 2: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Summary of Visual Redness at day 31; Test type: Superiority; p = 0.392, ANCOVA; Mean Difference (Final Values) = -0.089, 95% CI 2-sided [-0.292 to 0.115]
Statistical Analysis 3: Comparison: Test Cream (2% Urea/20% Glycerol) vs Reference Cream 2: Diprobase® Cream (Cream Without Humectants); Summary of Visual Redness at day 31; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.447, 95% CI 2-sided [-0.652 to -0.242]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout duration of the study, i.e. from day 1 to day 31
Description: Treatment emergent AEs were defined to be those starting on or after visit 1 treatment dispensing, or those without an onset date.
Groups:
- Test Cream (2% Urea/20% Glycerol); Reference Cream 1: Miniderm® 20% Cream (20% Glycerol); Reference Cream 2: Diprobase® Cream (Cream Without Humectants): 1 Finger Tip Unit of cream was applied to 1 of 4 skin areas on the lower volar forearm of the participant every morning and evening for 28 days
- Untreated: 1 of 4 skin areas on the lower volar forearm of the participant was left untreated
Arm/Group | Test Cream (2% Urea/20% Glycerol) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) | Untreated
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 1/49 | 6/49 | 15/49 | 0/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Cream (2% Urea/20% Glycerol) (N=49) | Reference Cream 1: Miniderm® 20% Cream (20% Glycerol) (N=49) | Reference Cream 2: Diprobase® Cream (Cream Without Humectants) (N=49) | Untreated (N=49)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Application site bruise (General disorders) | 0 | 0 | 2 | 0
Application site eczema (General disorders) | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 0 | 1 | 3 | 0
Application site papules (General disorders) | 0 | 2 | 0 | 0
Application site pruritus (General disorders) | 0 | 0 | 2 | 0
Application site rash (General disorders) | 0 | 0 | 3 | 0
Application site reaction (General disorders) | 0 | 0 | 1 | 0
Application site urticaria (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clause 10 of the Clinical Trial Agreement:

The Sponsor agrees that the Principal Investigator shall be permitted to present at symposia, national and regional professional meetings and to publish in journals, theses or dissertations, or otherwise of their own choosing, the methods and Results of the Clinical Trial, subject to this Clause 10 and any publication policy described in the Protocol, provided any such policy is consistent with the Joint Position.

DOCUMENTS (2):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT03901144/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT03901144/SAP_001.pdf